Preventing Sexual Violence Through a Comprehensive, Peer-led Initiative

NCT03207386

August 19, 2021

## **Study Protocol**

Written parental consent and student assent were required for youth to complete the study, consisting of five survey waves. Any youth in grades 7 to 10 (n = 4,172) at the beginning of the Fall 2017 semester were eligible and invited to enroll in the survey; the first survey occurred between October 2017 and December 2017. We used intensive recruitment procedures such that the consent forms were sent to parents in multiple ways (i.e., via their students from school, mailings, email) and we called and conducted home visits to households in which consent forms had not been returned. We also had multiple ways in which the consent forms could be returned (e.g., email, text, in person). At study initiation, of the 4,172 eligible students, the majority (n = 3,257; 78.0%) of youth returned the consent forms, and of those that returned the forms the majority (n = 2,667; 81.8%) of guardians gave permission for their student to take the survey. Most students (n = 2,232; 83.6%) with guardian permission took the survey. Figure 1 depicts eligibility and participation by wave. Past W1, we conducted ongoing study recruitment, such that we mailed consent forms to new students and followed up with calls and home visits, provided consent forms during in-school surveys, and offered consent forms at various community and school events.

The survey was administered on computers in school by trained research staff. All students had unique logins that were created in part so that students only with parental permission could access the survey. Students received a small incentive (e.g., fruit snack, pencil) and were entered to win one of twenty \$100 gift cards which increased by \$50 at each of the four subsequent surveys. Students who completed all surveys were entered into a drawing to receive a large prize equal to \$1,000 (e.g., tablets, pizza party). At each wave, students who missed the inschool survey (n = 475-1,289 across waves), were sent a letter in the mail requesting that they

take the survey online; instructions were provided for how to take the survey online. Return rate of these out-of-school surveys ranged from 1.8% to 8.4%. Overall, retention from W1 ranged from 58.3% to 85.6% across waves. The highly transient nature of the community where data were collected was a large factor in participant attrition; the most common reason for not participating was absence from school, and many of those absences were from students who had left the district. If students who left the district were not considered in retention analysis (e.g., removed from the denominator), retention from W1 ranged from 87.9% to 98.7%. We identified inattentive responders (students taking the survey) using questions like "Do you have more than 10 kids?" By the last wave, 108 participants (4.1%) were identified as an inattentive responder and removed from analyses.